CLINICAL TRIAL: NCT07315022
Title: Enhanced Recovery After Surgery-Based Multimodal Preemptive Analgesia for Perioperative Management in Transarterial Chemoembolization of Intermediate-to-Advanced Hepatocellular Carcinoma: a Multicenter Retrospective Cohort Study
Brief Title: Enhanced Recovery After Surgery-Based Multimodal Preemptive Analgesia for Perioperative Management in Transarterial Chemoembolization of Intermediate-to-Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangzhou Institute of Cancer Reasearch, the Affiliated Cancer Hospital, Guangzhou Medical University (Unknown); Jinshazhou Hospital of Guangzhou University of Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Jiaping Li, Chief Physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMAT2025
Record Dates: First submitted 2025-12-05; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Enhanced Recovery After Surgery; Multimodal Analgesia; Real-world Study; Transarterial Chemoembolization
Keywords: Enhanced Recovery After Surgery; Hepatocellular Carcinoma; Transarterial Chemoembolization; Multimodal Analgesia; Real-World Study; Hydromorphone; Flurbiprofen axetil
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hydromorphone; flurbiprofen axetil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A:hydromorphone + flurbiprofen axetil (Experimental): Group A received hydromorphone hydrochloride combined with flurbiprofen axetil via PCIA. Hydromorphone hydrochloride 6 mg (2 mL:2 mg, Hubei Yichang Humanwell Pharmaceutical) + flurbiprofen axetil 50 mg (5 mL:50 mg, Beijing Tide Pharmaceutical) were diluted with normal saline to 100 ml and loaded into a PCIA pump (48-h cycle). The pump was initiated 15 min before surgery, with settings of background infusion 2 ml/h, bolus dose 2 ml, and lockout interval 15 min. Patients could self-administer boluses when the numerical pain rating scale (NRS) score was ≥4, with repeated presses during lockout having no effect. For patients with an NRS score ≥4 after two effective boluses, hydromorphone 1 mg diluted in normal saline to 10 ml was administered as a slow push over 2-3 min.
  Interventions: Drug: hydrochloride hydromorphone + flurbiprofen axetil
- conventional analgesia (Active Comparator): Group B received on-demand analgesia. When the NRS score was ≥4, flurbiprofen axetil 50 mg was administered intravenously, with intramuscular tramadol 100 mg added if analgesia was inadequate.
  Interventions: Drug: conventional analgesia

INTERVENTIONS:
Drug: hydrochloride hydromorphone + flurbiprofen axetil — Group A received hydromorphone hydrochloride combined with flurbiprofen axetil via PCIA. The pump was initiated 15 min before surgery, with settings of background infusion 2 ml/h, bolus dose 2 ml, and lockout interval 15 min.
  Arms: A:hydromorphone + flurbiprofen axetil
Drug: conventional analgesia — When the NRS score was ≥4, flurbiprofen axetil 50 mg was administered intravenously, with intramuscular tramadol 100 mg added if analgesia was inadequate.
  Arms: conventional analgesia

SUMMARY:
To evaluate the effectiveness of the combination of hydrochloride hydromorphone and flurbiprofen ester for post-TACE intravenous patient-controlled intravenous analgesia (PCIA).

DETAILED DESCRIPTION:
This multicenter retrospective study analyzed clinical data from 129 patients with intermediate or advanced HCC who underwent TACE at three centers. Patients were divided into perioperative analgesia protocol groups: Group A (n=85) received patient-controlled intravenous analgesia-based multimodal preemptive analgesia (hydromorphone hydrochloride 6 mg, flurbiprofen axetil 50 mg) with background infusion. Group B (n=44) received conventional on-demand analgesia (intraoperative intravenous flurbiprofen axetil 50 mg, intramuscular tramadol 100 mg as needed for pain). Outcome measures included numerical rating pain scale scores, perioperative adverse events, inflammatory markers, hepatic function indicators, analgesia satisfaction, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or clinically diagnosed with hepatocellular carcinoma according to the "Guidelines for Diagnosis and Treatment of Primary Liver Cancer" issued by the National Health Commission of China in 2024;
2. staged as China Liver Cancer Stage II-III1 or 2022 Barcelona Clinic Liver Cancer stage B-C14;
3. liver function classified as Child-Pugh grade A or B;
4. ECOG PS score 0-215;
5. meeting the following hematological criteria: white blood cell count ≥3×10⁹/L, platelet count ≥50×10⁹/L, hemoglobin ≥80 g/L, serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤twice the upper limit of normal (ULN), serum creatinine ≤1.5×ULN, INR <1.5 or prothrombin time <ULN + 4 s, albumin (ALB) ≥30 g/L, total bilirubin <34 mmol/L.

Exclusion Criteria:

1. History of iodine contrast allergy;
2. severe psychological or psychiatric disorders;
3. history of long-term analgesic medication use;
4. severe cardiopulmonary disease;
5. severe uncontrolled infection;
6. incomplete medical records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Perioperative numerical pain rating scale (NRS) score | From the start of the operation to 24 hours after the operation
  The NRS was used to assess pain intensity intraoperatively, immediately postoperatively, and at 1 h, 4 h, 8 h, 12 h, and 24 h postoperatively, with scores ranging 0-10 (0=no pain, 1-3=mild pain, 4-6=moderate pain, 7-10=severe pain).

SECONDARY OUTCOMES:
Surgical Duration | From the start of the operation to the end of the operation
  Total time from puncture initiation to completion of dressing (min).
Adverse Events | From the start of the operation to 24 hours after the operation
  Adverse events within 24 h postoperatively were recorded, including elevated ALBI scores, ALT and AST >2×ULN, nausea and vomiting, drowsiness and dizziness, pruritus, and urinary difficulty, with related indicator changes and incidence documented.
Analgesia Satisfaction | At 24 hours postoperatively
  At 24 h postoperatively, patients' subjective experiences were assessed using a 5-point Likert scale (5=very satisfied, 4=satisfied, 3=neutral, 2=dissatisfied, 1=very dissatisfied).
Cost-Effectiveness Analysis | From the start of the operation to the end of perioperative period
  TACE perioperative analgesia costs plus postoperative hospitalization costs were used as the cost indicator (C), with analgesia satisfaction ≥4 as the effectiveness indicator (E). The average cost approach was used for incremental cost-effectiveness analysis (ΔC/ΔE).

OTHER OUTCOMES:
Serum Inflammatory Markers | preoperatively and on the second postoperative morning
  Fasting venous blood was collected preoperatively and on the second postoperative morning to measure procalcitonin (PCT)(ng/ml) and interleukin-6 (IL-6)(pg/ml) levels.
Hepatic Function Indicators | preoperatively and on the second postoperative morning
  Fasting venous blood was collected preoperatively and on the second postoperative morning to measure serum alanine aminotransferase (ALT)(U/L), aspartate aminotransferase (AST)(U/L), albumin (ALB)(g/L), total bilirubin levels(μmol/L), and ALB-bilirubin (ALBI) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Result] Thompson AR, Vernamonti JP, Rollins P, Speck KE. Implementing Change: Sustaining Enhanced Recovery After Surgery Protocols in Pediatric Surgery Using Iterative Assessments. J Surg Res. 2024 Jun;298:371-378. doi: 10.1016/j.jss.2024.03.039. Epub 2024 Apr 25. PMID 38669783
- [Result] Ribero L, Santia MC, Borchardt K, Zabaneh F, Beck A, Sadhu A, Edwards K, Harrelson M, Pinales-Rodriguez A, Yates EM, Ramirez PT. Surgical site infection prevention bundle in gynecology oncology surgery: a key element in the implementation of an enhanced recovery after surgery (ERAS) program. Int J Gynecol Cancer. 2024 Sep 2;34(9):1445-1453. doi: 10.1136/ijgc-2024-005423. PMID 38876786
- [Result] Zhou J, Sun H, Wang Z, Cong W, Zeng M, Zhou W, Liu L, Wen T, Kuang M, Zhang B, Tao K, Han G, Yan Z, Wang M, Liu R, Guo J, Zeng Z, Liang P, Ren Z, Hou J, Zhang Y, Liu X, Pan H, Bi F, Liang C, Chen M, Yan F, Xu H, Xie X, Ju S, Ji Y, Yun J, Li Z, Bai X, Cai D, Chen W, Chen Y, Chen Y, Cheng W, Cheng S, Dai Z, Dai C, Gao Q, Guo R, Guo W, Guo Y, Hua B, Huang X, Jiang H, Jia W, Li Q, Li T, Li X, Li X, Li Y, Li Y, Liang J, Liang X, Ling C, Liu H, Liu T, Lu S, Lv G, Mao Y, Meng Z, Peng T, Ren W, Shi G, Shi H, Shi M, Song T, Tan G, Wang J, Wang K, Wang L, Wang W, Wang X, Wang Z, Xiang B, Xia J, Xing B, Xu J, Xu J, Yang J, Yang X, Yang Y, Yang Y, Yao X, Yin Z, Yuan Z, Zeng Y, Zeng Y, Zhang B, Zhang L, Zhang S, Zhang T, Zhang Z, Zhao M, Zhao Y, Zheng H, Zhou L, Zhu J, Zhu K, Shi Y, Liu R, Zhang L, Xiao Y, Yang C, Wu Z, Ding Z, Zhu X, Tang Z, Huang X, Han H, Wu H, Chen M, Wang W, Li Q, Cai J, Shen F, Cai X, Qin S, Teng G, Fan J. China Liver Cancer Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2024 Edition). Liver Cancer. 2025 Jul 10;14(6):779-835. doi: 10.1159/000546574. eCollection 2025 Dec. PMID 41063733
- [Result] Liu J, Zhang W, Lu H, Li H, Zhou X, Li J, Han X. Drug-eluting bead trans-arterial chemoembolization combined with microwave ablation therapy vs. microwave ablation alone for early stage hepatocellular carcinoma: a preliminary investigation of clinical value. J Cancer Res Clin Oncol. 2022 Jul;148(7):1781-1788. doi: 10.1007/s00432-021-03760-x. Epub 2021 Aug 17. PMID 34405295
- [Result] Zhu XD, Li KS, Sun HC. Adjuvant therapies after curative treatments for hepatocellular carcinoma: Current status and prospects. Genes Dis. 2020 Feb 29;7(3):359-369. doi: 10.1016/j.gendis.2020.02.002. eCollection 2020 Sep. PMID 32884990
- [Result] Jones DB, Abu-Nuwar MRA, Ku CM, Berk LS, Trainor LS, Jones SB. Less pain and earlier discharge after implementation of a multidisciplinary enhanced recovery after surgery (ERAS) protocol for laparoscopic sleeve gastrectomy. Surg Endosc. 2020 Dec;34(12):5574-5582. doi: 10.1007/s00464-019-07358-w. Epub 2020 Jan 14. PMID 31938928
- [Result] Interventional perioperative committee of Chinese College of Interventionalists, clinical practice guideline committee of Chinese college of interventionalists. Expert consensus on perioperative pain management for interventional treatment of hepatic malignancies (2022). J Interv Radiol. 2022;31(10):943-948.
- [Result] Meyer T, Fox R, Ma YT, Ross PJ, James MW, Sturgess R, Stubbs C, Stocken DD, Wall L, Watkinson A, Hacking N, Evans TRJ, Collins P, Hubner RA, Cunningham D, Primrose JN, Johnson PJ, Palmer DH. Sorafenib in combination with transarterial chemoembolisation in patients with unresectable hepatocellular carcinoma (TACE 2): a randomised placebo-controlled, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2017 Aug;2(8):565-575. doi: 10.1016/S2468-1253(17)30156-5. Epub 2017 Jun 23. PMID 28648803
- [Result] Golfieri R, Giampalma E, Renzulli M, Cioni R, Bargellini I, Bartolozzi C, Breatta AD, Gandini G, Nani R, Gasparini D, Cucchetti A, Bolondi L, Trevisani F; PRECISION ITALIA STUDY GROUP. Randomised controlled trial of doxorubicin-eluting beads vs conventional chemoembolisation for hepatocellular carcinoma. Br J Cancer. 2014 Jul 15;111(2):255-64. doi: 10.1038/bjc.2014.199. Epub 2014 Jun 17. PMID 24937669
- [Result] Benzakoun J, Ronot M, Lagadec M, Allaham W, Garcia Alba C, Sibert A, Vilgrain V. Risks factors for severe pain after selective liver transarterial chemoembolization. Liver Int. 2017 Apr;37(4):583-591. doi: 10.1111/liv.13235. Epub 2016 Sep 2. PMID 27529160
- [Result] Zhou B, Wang J, Yan Z, Shi P, Kan Z. Liver cancer: effects, safety, and cost-effectiveness of controlled-release oxycodone for pain control after TACE. Radiology. 2012 Mar;262(3):1014-21. doi: 10.1148/radiol.11110552. PMID 22357901